CLINICAL TRIAL: NCT05616689
Title: Bundled Hyperpolypharmacy Deprescribing: Implementation and Evaluation of a System-wide Quality Improvement Intervention
Brief Title: Bundled Hyperpolypharmacy Deprescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RDO KPNC 20 - 008
Record Dates: First submitted 2022-10-19; First posted 2022-11-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Polypharmacy
Keywords: deprescribing; polypharmacy; drug safety; randomized controlled trial; pharmacist; shared decision making; optimal prescribing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bundled hyperpolypharmacy intervention (Experimental): Eligible participants with physician authorization who are randomly assigned to intervention
  Interventions: Other: Bundled hyperpolypharmacy
- Control (No Intervention): Eligible participants with physician authorization who are randomly assigned to usual care

INTERVENTIONS:
Other: Bundled hyperpolypharmacy — Bundled hyperpolypharmacy playbook to be used by pharmacist, with physician approval, in shared decision making with participant,
  Arms: Bundled hyperpolypharmacy intervention

SUMMARY:
Older patients using many prescription drugs (hyperpolypharmacy) may be at increased risk of adverse drug effects. This randomized controlled trial tested the effectiveness and safety of a quality intervention intended to reduce hyperpolypharmacy. The study was set at Kaiser Permanente Northern California, an integrated health system with multiple pre-existing deprescribing workflows. Eligible patients were aged ≥76 years using ≥10 prescription medications. The intervention included physician-pharmacist collaborative drug therapy management, standard-of-care practice recommendations, shared decision-making, and deprescribing protocols administered by telephone over multiple cycles for a maximum of 180 days after allocation. A priori primary effectiveness endpoints included change in the number of medications and in the prevalence of geriatric syndrome from 181-365 days after allocation. Second endpoints included utilization and adverse drug withdrawal effects. Information was obtained from the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente patients
* Age ≥76 years
* ≥10 drugs (excluding topicals) where

  * drug filled ≥2 times in the past year and
  * drug last filled < 180 days ago

Exclusion Criteria:

* less than 12 months preceding enrollment at Kaiser Permanente
* no primary care practitioner assigned
* on dialysis
* history of heart, liver, lung, breast, or bone marrow transplant
* in hospice
* under active treatment for cancer during the past 12 months
* has received an intervention through the Pharmacy Targeted Deprescribing Program in the preceding year.

Min Age: 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2471 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of geriatric syndrome | Difference between (days 181-365 after randomization) and (180 days before randomization)
  Change in prevalence for any of the following: Falls (hip fracture, lower leg fracture, osteoporosis with fracture, pathologic fracture, osteonecrosis; gait; repeated falls; syncope; tripping; reduced mobility), Cognition (Somnolence; awareness; dizziness; malaise; Urinary incontinence (Unspecified urinary incontinence; retention of urine, unspecified; functional urinary incontinence; stress incontinence ; other specified urinary incontinence) and Pain (Drug induced headache; joint pain; muscle weakness, rhabdomyolysis, spas; myalgia)
Change in number of medications | Difference between (days 181-365 after randomization) and (180 days before randomization)
  Change in number of dispensed medications recorded in the comprehensive, integrated pharmacy information system

SECONDARY OUTCOMES:
Utilization | Difference between (days 181-365 after randomization) and (180 days before randomization)
  Change in number of outpatient visits, inpatient visits, and emergency department visits.

OTHER OUTCOMES:
Adverse drug withdrawal effects | Difference between (days 181-365 after randomization) and (180 days before randomization)
  Change in prevalence of lower respiratory, cardiovascular, gastrointestinal, hyperuricemia, and elevated blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Herrinton, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herrinton LJ, Lo K, Alavi M, Alexeeff SE, Butler KM, Chang C, Chang CC, Chu VL, Krishnaswami A, Deguzman LH, Prausnitz S, Mason MD, Draves M. Effectiveness of Bundled Hyperpolypharmacy Deprescribing Compared With Usual Care Among Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2322505. doi: 10.1001/jamanetworkopen.2023.22505. PMID 37428504